CLINICAL TRIAL: NCT04802226
Title: Optimization of the Self-exclusion Procedure
Acronym: OSE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Local /2020/AL
Record Dates: First submitted 2021-03-11; First posted 2021-03-17 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Sports Betting Players

STUDY DESIGN:
Intervention Model Description: Naturalistic randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- optimized self-exclusion procedure A (Experimental): optimized self-exclusion procedure including content optimization with brief intervention, normative feedback, motivational approach, a personal story of a peer who had a positive experience using the tool, re-contact before the end of the self-exclusion period to propose an extension of the period outside the gambling plateform
  Interventions: Other: self exclusion procedure
- standard self-exclusion B (Other): standard self-exclusion with a single neutral notification email
  Interventions: Other: self exclusion procedure

INTERVENTIONS:
Other: self exclusion procedure — self exclusion procedure( responsible gambling tool)

SUMMARY:
It has been shown that self-excluded gamblers are very heavy gamblers, and that it is not possible to distinguish between those who report self-exclusion for addictive reasons and those who self-exclude for commercial reasons, which strongly suggests that all self-excluded people are "self-diagnosed" problem gamblers. Several studies converge in recognizing self-excluded people as problem gamblers who have lost control of their gambling and are seeking to protect themselves by taking action, self-exclusion, to change their behaviour and protect themselves.

Several reviews of the literature on interventions for problem gamblers have recently identified self-exclusion as an intervention for problem gamblers.

However, the effectiveness of the current self-exclusion system appears to be limited, particularly for short self-exclusions and for heavier gamblers.

Considering that self-exclusion is an intervention for and by people who have developed a gambling disorder, it currently consists exclusively of a behavioural intervention, in the sense that it prevents the behaviour. It would then be possible to optimize this intervention by enriching it with other components that have been shown to be effective with problem gamblers or in other addictions: a brief intervention including a motivational, cognitive approach, personalized normative feedback, referral to online help services (cresus and gambling infoservice), and repeated contact to suggest an extension of the self-exclusion period without having to return to the gambling environment. We hypothesize improved efficacy as measured by reduced gambling for longer after an initial optimized self-exclusion compared to self-exclusion with the standard procedure. Days will be randomized according to an a priori randomization list, not players.

DETAILED DESCRIPTION:
Main Objective:

The primary objective of the study is to evaluate the effect of the optimized self-exclusion procedure, compared to the existing procedure, on the intensity of gambling.

- Primary endpoint The primary endpoint is the change in total net loss over the last 4 weeks, between the last 4 weeks prior to self-exclusion T0, and the last 4 weeks at 12 months T2.

2.2 Secondary objectives The secondary objectives of the study are to assess early effect at 6 months and maintenance of effect at 18 months.

- Secondary endpoints:

The secondary objectives of the study are to evaluate early efficacy at 6 months and maintenance of efficacy at 18 months. The endpoint used is the change in total net loss over the last 4 weeks, between the last 4 weeks prior to self-exclusion, and the last 4 weeks at 6 T1 and 18 months T3. The other criteria will be the change between T0 and T1,2, and 3 of the following variables (total of the last 4 weeks unless otherwise specified):

* Total deposit
* Total bet per game
* Compulsiveness (as defined by three consecutive deposits in a 12-hour period) (yes/no) (number of episodes)
* Maximum number of deposits within one hour of a bet,
* Total loss per game (average)
* Number of gambling sessions (all games) in a clinical sense; session is defined as the gambling behavior itself; we will consider the beginning of a session when a gambling action occurs after no gambling action has occurred for at least 30 minutes, and the end of the gambling session a gambling action followed by no gambling action for 30 minutes.
* Session duration (average)
* Total playing time defined as the sum of the session durations
* Extension of self-exclusion (yes no)
* Second and subsequent self-exclusion (yes no, number)
* Exceeding 80% moderators (sum).

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Must be self-exclude for the first time
* Must be Online sports betting player
* Must be self-exclusion of 3 months or less (minimum 3 days)

Exclusion Criteria:

* Player who has objected to the use of his collected data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2554 (Actual)
Dates: Start 2021-01-02 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
change in total net loss over the last 4 weeks, between the last 4 weeks prior to self-exclusion T0, and the last 4 weeks at 12 months T2 | between the last 4 weeks before self-exclusion T0, and the last 4 weeks at 12 months T2

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nîmes, Nîmes, France

IPD SHARING:
Plan to Share IPD: No